CLINICAL TRIAL: NCT03352336
Title: A Comparison Between Two Methods for Estimating the Extent of Perioperative Atelectasis
Brief Title: Estimation of Perioperative Atelectasis
Status: Completed | Type: Observational
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Edmark, Principal Investigator, Region Västmanland
Other Study IDs: Dnr 2017/27:2
Record Dates: First submitted 2017-11-19; First posted 2017-11-24 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Atelectasis; Oxygenation
Keywords: Atelectasis; Oxygenation; Venous admixture; Computed Tomography; Oxygenation test
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood gases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will compare an oxygenation test based on arterial blood gas analysis with computed tomography for estimating the extent of atelectasis.

DETAILED DESCRIPTION:
Computed tomography of the lungs is the gold standard for investigating the extent of atelectasis, which is common in the perioperative setting. Atelectasis increase the risk of postoperative pulmonary complications and result in pulmonary shunt, which is one of the two major causes of impaired oxygenation. The other cause is admixture of venous blood from poorly ventilated regions of the lungs. The investigators have developed an oxygenation test utilizing arterial blood gas analysis at different inspired fractions of oxygen, which may be used to distinguish between these two causes. This observational study aims to establish the agreement between computed tomography and the oxygenation test for estimating the extent of atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class I-II.
* Non-abdominal day case surgery under general anesthesia.
* Patients enrolled in study registered in ClinicalTrials with NCT ID.

Exclusion Criteria:

* Arterial oxygen saturation (SpO2) <90 % with 40% Venturi mask.
* Unstable postoperative condition needing immediate treatment.

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling inclusion and exclusion criteria while attending the day case department of Köping county hospital in Region Västmanland.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Atelectasis area | 30 min after emergence from anesthesia
  Atelectasis area as studied by computed tomography

SECONDARY OUTCOMES:
Pulmonary shunt estimated by a standardised oxygenation test | 30 min after emergence from anesthesia
  Pulmonary shunt estimated by a standardised oxygenation test using

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Edmark, M.D., Ph.D., Study Director — Region Västmanland
Locations (1):
- Västmanlands sjukhus Köping, Köping, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome will be available.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the board of the local clinical research center in Region Vastmanland. Requestors will be required to sign a Data Access Agreement.